CLINICAL TRIAL: NCT02219516
Title: A Phase 1, Single-Dose, Open Label, Pharmacokinetic and Pharmacodynamic Study of RDEA3170 in Adult Male Subjects With Mild, Moderate, and Severe Renal Impairment
Brief Title: Mild, Moderate and Severe Renal Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA3170-108
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — verinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1: Mild renal impairment (Experimental): RDEA3170 15 mg once daily fasted
  Interventions: Drug: RDEA3170
- Cohort 2: Moderate renal impairment (Experimental): RDEA3170 15 mg once daily fasted
  Interventions: Drug: RDEA3170
- Cohort 3: Severe renal impairment (Experimental): RDEA3170 15 mg once daily fasted
  Interventions: Drug: RDEA3170
- Cohort 4: Control subjects with normal renal function (Experimental): RDEA3170 15 mg once daily fasted
  Interventions: Drug: RDEA3170

INTERVENTIONS:
Drug: RDEA3170

SUMMARY:
This is a Phase 1, single-dose, open-label, pharmacokinetic (PK) and pharmacodynamic (PD) study of RDEA3170 in adult male subjects with mild, moderate, and severe renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body weight ≥ 50 kg (110 lbs.) and a body mass index ≥ 18 and ≤ 40 kg/m2.
* Subject with renal impairment, as determined at Screening, with creatinine clearance as calculated by the Cockcroft-Gault formula of 60 to < 90 mL/min (mild impairment), 30 to < 60 mL/min (moderate impairment), or 15 to < 30 mL/min (severe impairment), or a matched control subject (by age and body mass index) with a creatinine clearance of ≥ 90 mL/min.
* Subject has a Screening serum urate level ≥ 4.5 mg/dL and ≤ 10 mg/dL

Exclusion Criteria:

* Subject has a history or clinical manifestations of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urological, or psychiatric disorders.
* Subject has a history or suspicion of kidney stones.
* Subject has a history of asthma.
* Subject has undergone major surgery within 3 months prior to Day 1.
* Subject has donated blood or experienced significant blood loss (> 450 mL) within 12 weeks prior to Day 1 or gave a plasma donation

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2016-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Hall, MD, Study Director — Ardea Biosciences, Inc.
Locations (4):
- United States (4):
  - Lakewood, Colorado
  - Orlando, Florida
  - Minneapolis, Minnesota
  - Knoxville, Tennessee

REFERENCES:
- [Derived] Smith WB, Hall J, Berg JK, Kazimir M, Yamamoto A, Walker S, Lee CA, Shen Z, Wilson DM, Zhou D, Gillen M, Marbury TC. Effect of Renal Impairment on the Pharmacokinetics and Pharmacodynamics of Verinurad, a Selective Uric Acid Reabsorption Inhibitor. Clin Drug Investig. 2018 Aug;38(8):703-713. doi: 10.1007/s40261-018-0652-2. PMID 29949102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 subjects were randomized
Pre-assignment Details: Thirty-one subjects were randomized to 1 of 4 cohorts. Cohort 1: mild renal impairment; Cohort 2: moderate renal impairment; Cohort 3: severe renal impairment and Cohort 4: normal renal function. All 31 subjects received a single dose of 15 mg RDEA3170 (6 x 2.5 mg) in the fasted state.
Groups:
- Cohort 1: Mild Renal Impairment + RDEA3170 15 mg: Mild Renal Impairment (eCrCl of 60 to < 90 mL/min) + RDEA3170 15 mg once daily (qd) fasted
- Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg: Moderate Renal Impairment (eCrCl of 30 to < 60 mL/min) + RDEA3170 15 mg qd fasted
- Cohort 3: Severe Renal Impairment + RDEA3170 15 mg: Severe Renal Impairment (eCrCl of 15 to < 30 mL/min) + RDEA3170 15 mg qd fasted
- Cohort 4: Normal Renal Function + RDEA3170 15 mg: Control subjects With Normal Renal Function (eCrCl of ≥ 90 mL/min) + RDEA3170 15 mg qd fasted
Period: Overall Study
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Started | 8 | 8 | 7 | 8
Completed | 8 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg | Total
Number analyzed (Participants) | 8 | 8 | 7 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63 (6.4) | 67 (14.9) | 58 (11.1) | 56 (4.7) | 61 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 7 | 8 | 31
Region of Enrollment [Number; unit: Participants]
  United States | 8 | 8 | 7 | 8 | 31

OUTCOME MEASURES:

1. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Time Frame: 5 weeks
Measure: Number; unit: Number of participants
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Number analyzed (Participants) | 8 | 8 | 7 | 8
Number of participants | 3 | 1 | 2 | 1

2. Secondary Outcome: Pharmacodynamics (PD) Profiles of Uric Acid From Serum and Urine
Time Frame: Screening, Day -1 ( -24, -21, -18, -and -12 hours predose), and Day 1 (within 30 minutes prior to dosing and at 3, 6, 12, 24, 30, 36, 48, 54, 60, and 72 hours postdose)
Measure: Mean (Standard Error); unit: Maximum Percentage (%) Change
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Number analyzed (Participants) | 8 | 8 | 7 | 8
Maximum Percentage (%) Change
  Serum Urate Maximum % Change | -36.9 (4.79) | -20.5 (2.62) | -12.6 (2.62) | -38.3 (5.24)
  Urine Uric Acid % Change (0-24h) | 118 (25.3) | 69.3 (19.0) | 72.5 (17.1) | 85.2 (15.2)
  Renal Clearance of Uric Acid % Change (0-24h) | 222 (50.5) | 96.7 (11.9) | 82.9 (16.6) | 163 (30.1)
  Fract. Excretion of Uric Acid % Change (0-24h) | 206 (44.9) | 89.6 (24.1) | 54.5 (17.0) | 159 (28.7)
  Urine Uric Acid % Change (24-48h) | -9.49 (6.68) | 4.18 (9.89) | 28.3 (11.2) | -1.54 (12.1)
  Urine Uric Acid % Change (48-72h) | -23.1 (7.63) | -16.0 (11.5) | 6.02 (20.2) | -20.8 (9.65)
  Renal Clearance of Uric Acid % Change (24-48h) | 42.1 (12.9) | 25.4 (9.40) | 34.5 (9.17) | 31.9 (16.8)
  Renal Clearance of Uric Acid % Change (48-72h) | 2.39 (6.84) | -0.439 (11.9) | 9.38 (21.5) | -8.12 (12.2)
  Fract. Excretion of Uric Acid % Change (24-48h) | 39.2 (10.8) | 28.7 (7.91) | 19.0 (4.89) | 27.8 (9.74)
  Fract. Excretion of Uric Acid % Change (48-72h) | 14.2 (9.43) | 4.18 (10.7) | 1.67 (4.01) | 2.27 (8.29)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax following a single administration of RDEA3170 to subjects with various degrees of renal function
Time Frame: Day 1: within 30 minutes prior to dosing and at 30 minutes, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 30, 36, 48, 54, 60, and 72 hours postdose
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Number analyzed (Participants) | 8 | 8 | 7 | 8
ng/mL | 25.6 [20.0 to 32.9] | 29.0 [22.8 to 37.0] | 38.2 [24.0 to 60.8] | 16.7 [12.6 to 22.3]
Statistical Analysis 1: Comparison: Cohort 1: Mild Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; Treatment as a fixed effect was used to analyze the natural log-transformed PK parameters and GLSMRs are back-transformed to the original scale; Geometric Least Squares Mean Ratio (%) = 153, 90% CI 2-sided [115 to 203]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 173, 90% CI 2-sided [131 to 230]
Statistical Analysis 3: Comparison: Cohort 3: Severe Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 228, 90% CI 2-sided [155 to 336]

4. Primary Outcome: Time of Occurrence of Maximum Observed Concentration (Tmax)
Description: Tmax following a single administration of RDEA3170 to subjects with various degrees of renal function
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Number analyzed (Participants) | 8 | 8 | 7 | 8
hr | 2.50 [1.00 to 4.00] | 3.00 [1.50 to 5.00] | 2.00 [1.50 to 4.00] | 2.50 [0.500 to 4.00]

5. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Sampling Timepoint (AUC Last)
Description: AUC last following a single administration of RDEA3170 to subjects with various degrees of renal function
Time Frame: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ng.hr/mL
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Number analyzed (Participants) | 8 | 8 | 7 | 8
ng.hr/mL | 197 [142 to 273] | 333 [246 to 451] | 316 [179 to 559] | 150 [123 to 182]
Statistical Analysis 1: Comparison: Cohort 1: Mild Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 131, 90% CI 2-sided [98.6 to 174]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 222, 90% CI 2-sided [171 to 287]
Statistical Analysis 3: Comparison: Cohort 3: Severe Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 211, 90% CI 2-sided [139 to 319]

6. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC∞)
Description: AUC∞ following a single administration of RDEA3170 to subjects with various degrees of renal function
Time Frame: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ng.hr/mL
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Number analyzed (Participants) | 8 | 8 | 7 | 8
ng.hr/mL | 201 [144 to 279] | 402 [225 to 634] | 372 [209 to 663] | 162 [120 to 218]
Statistical Analysis 1: Comparison: Cohort 1: Mild Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 124, 90% CI 2-sided [88.8 to 173]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 248, 90% CI 2-sided [168 to 366]
Statistical Analysis 3: Comparison: Cohort 3: Severe Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 230, 90% CI 2-sided [146 to 363]

7. Primary Outcome: Apparent Terminal Half-life (t1/2)
Description: t1/2 following a single administration of RDEA3170 to subjects with various degrees of renal function
Time Frame: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Number analyzed (Participants) | 8 | 8 | 7 | 8
hr | 9.53 [7.42 to 12.2] | 20.6 [9.96 to 42.4] | 22.0 [14.2 to 34.1] | 13.0 [7.91 to 21.5]

8. Primary Outcome: Non-renal Clearance From Time 0 to 72 Hours Postdose (CLNR 0-72)
Description: CLNR 0-72 following a single administration of RDEA3170 to subjects with various degrees of renal function
Time Frame: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Number analyzed (Participants) | 8 | 8 | 7 | 8
L/hr | 74.9 [53.9 to 104] | 44.5 [33.0 to 59.9] | 47.2 [26.6 to 83.5] | 98.6 [80.9 to 120]
Statistical Analysis 1: Comparison: Cohort 1: Mild Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 76.0, 90% CI 2-sided [57.1 to 101]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 45.1, 90% CI 2-sided [34.9 to 58.3]
Statistical Analysis 3: Comparison: Cohort 3: Severe Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 47.8, 90% CI 2-sided [31.5 to 72.5]

9. Primary Outcome: Total Body Clearance Corrected for Bioavailability (CL/F)
Description: CL/F following a single administration of RDEA3170 to subjects with various degrees of renal function
Time Frame: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Number analyzed (Participants) | 8 | 8 | 7 | 8
L/hr | 74.8 [53.7 to 104] | 37.3 [23.7 to 58.9] | 40.3 [22.6 to 71.7] | 92.6 [68.7 to 125]
Statistical Analysis 1: Comparison: Cohort 1: Mild Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 80.8, 90% CI 2-sided [57.9 to 113]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 40.3, 90% CI 2-sided [27.3 to 59.5]
Statistical Analysis 3: Comparison: Cohort 3: Severe Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 43.5, 90% CI 2-sided [27.5 to 68.7]

10. Primary Outcome: Renal Clearance Time 0 to 72 Hours Postdose (CLR 0-72)
Description: CLR 0-72 following a single administration of RDEA3170 to subjects with various degrees of renal function
Time Frame: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Number analyzed (Participants) | 8 | 8 | 7 | 8
mL/min | 12.9 [8.16 to 20.4] | 7.87 [3.36 to 18.4] | 2.86 [1.84 to 4.45] | 13.5 [9.03 to 20.2]
Statistical Analysis 1: Comparison: Cohort 1: Mild Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 95.4, 90% CI 2-sided [60.6 to 150]
Statistical Analysis 2: Comparison: Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 58.3, 90% CI 2-sided [30.2 to 113]
Statistical Analysis 3: Comparison: Cohort 3: Severe Renal Impairment + RDEA3170 15 mg vs Cohort 4: Normal Renal Function + RDEA3170 15 mg; Test type: Non-Inferiority or Equivalence — Informal BE assessment using the conventional BE limits of 80% to 125%; Fixed Effects Model; [statistical method as in outcome 3, analysis 1]; Geometric Least Squares Mean Ratio (%) = 21.2, 90% CI 2-sided [13.6 to 32.8]

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: Overall number of baseline participants used to determine number of participants at risk.
Arm/Group | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg | Cohort 4: Normal Renal Function + RDEA3170 15 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 1/8 | 2/7 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Mild Renal Impairment + RDEA3170 15 mg (N=8) | Cohort 2: Moderate Renal Impairment + RDEA3170 15 mg (N=8) | Cohort 3: Severe Renal Impairment + RDEA3170 15 mg (N=7) | Cohort 4: Normal Renal Function + RDEA3170 15 mg (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudofolliculitis barbae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.